CLINICAL TRIAL: NCT05276726
Title: A Phase Ib/II ,Single Arm, Multi-Center, Open Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Evidence of JAB-21822 in Advanced or Metastatic Non-small Cell Lung Cancer With a KRAS p.G12C and STK11 Co-mutation and Wild-type KEAP1
Brief Title: A Study of JAB-21822 in Advanced or Metastatic NSCLC With KRAS p.G12C and STK11 Co-mutation and Wild-type KEAP1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JAB-21822-1003
Record Dates: First submitted 2022-03-03; First posted 2022-03-11 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 1 ,Dose Exploration ,monotherapy (Experimental): Dose escalation of JAB21822 will be administered as monotherapy to determine the MTD and RP2D
  Interventions: Drug: JAB 21822
- Phase 2, Dose Expansion, Part1 monotherapy (Experimental): Part 1 dose expansion is to evaluate the safety and clinical activity of JAB-21822 at RP2D in subjects with previously untreated advanced non-small cell lung cancer (NSCLC)
  Interventions: Drug: JAB 21822
- Phase 2 Dose Expansion, Part 2 monotherapy (Experimental): Part 2 dose expansion is to evaluate the safety and clinical activity of JAB-21822 at RP2D in subjects who had received at least one previous line of systemic therapy for NSCLC
  Interventions: Drug: JAB 21822

INTERVENTIONS:
Drug: JAB 21822 — Administered orally

SUMMARY:
Evaluate the safety and tolerability, drug levels, and clinical activity of JAB-21822 in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) whose tumors with KRAS p.G12C mutation and a serine/threonine kinase 11 (STK11) co-mutation.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of JAB-21822 during Dose Escalation phase and preliminary antitumor activity in patients with NSCLC with concurrent KRAS G12C mutant and STK11 mutant and KEAP wild type either treatment naïve or at least one line prior therapy for advance disease during the expansion phase..

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically documented, locally-advanced or metastatic NSCLC with KRAS p.G12C mutation identified through molecular testing.
2. STK11 co-mutation and KEAP1 Wild-Type (local confirmation)
3. Treatment naïve or have received at least 1 prior standard therapy for advanced NSCLC
4. ECOG 0-1

Exclusion Criteria:

1. Has CNS metastases or carcinomatous meningitis, except treated CNS metastases with no evidence of radiographic progression or hemorrhage for at least 28 days
2. Any severe and/or uncontrolled medical conditions
3. Active infection requiring systemic treatment within 7 days
4. Therapeutic radiation therapy within 3 weeks of study day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation phase Number of participants with dose limiting toxicities (DLTs) | At the end of Cycle 1 (each cycle is 21 days)
  A DLT is defined as the clinically significant treatment-related adverse event or abnormal laboratory values assessment during the first 21 days of Cycle 1. It excludes adverse events (AEs) that are deemed clearly related to underlying disease, progression, or intercurrent illness.
Dose Escalation phase: Number of participants with adverse events | Up to 3 years
  Patients will be assessed for incidence and severity of AEs according to NCI-CTCAE 5.0 criteria
Dose Expansion phase: Objective response rate (ORR) | Up to 3 years - from baseline to confirmed Progressive Disease per RECIST.
  ORR is defined as the percentage of participants with complete response (CR) or partial response (PR) per RECIST v 1.1

SECONDARY OUTCOMES:
Dose Escalation phase: Objective response rate (ORR) | Up to 3 years - from baseline to RECIST confirmed Progressive Disease
  ORR is defined as the percentage of participants with complete response (CR) or partial response (PR) per RECIST v 1.1
Dose Escalation and Dose Expansion phase: Progression-free survival (PFS) | Up to 3 years
  PFS is defined as the interval of time between the date of first treatment to the earliest date of disease progression per RECIST1.1 or death whichever occurs first
Dose Escalation and Dose Expansion phase: Duration of response (DOR) | Up to 3 years
  DOR is defined as the time from the participant's initial objective response (CR or PR) to disease progression per RECIST v1.1 or death due to any cause, whichever occurs first.
Dose Escalation and Dose Expansion phase: Disease Control Rate (DCR) | Up to 3 years
  DCR is defined as percentage of participants with complete response (CR), partial response (PR), or stable disease (SD) per RECIST v1.1
Dose Escalation and Dose Expansion phase: Overall Survival (OS) | Up to 3 years
  Defined as time from first treatment to death by any cause
Dose Escalation and Dose Expansion phase: Time to response (TTR) | Up to 3 years
  Defined as time from first treatment to first evidence of PR or CR
Dose Expansion phase: Number of participants with adverse events | Up to 3 years
  Patients will be assessed for incidence and severity of adverse events (AEs) according to NCI-CTCAE criteria
Dose Escalation and Dose Expansion phase: Plasma concentration (Cmax) | Up to 3 Years
  Cmax of JAB-21822 will be measured by using plasma PK samples
Dose Escalation and Dose Expansion phase: Time to achieve Cmax (Tmax) | Up to 3 Years
  Tmax of JAB-21822 will be measured by using plasma PK samples
Escalation and Dose Expansion phase：Area under the plasma concentration-time curve (AUC) | Up to 3 Years
  AUC of JAB-21822 will be measured by using plasma PK samples

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - Research site08, Beijing, Beijing Municipality
  - Research site09, Beijing, Beijing Municipality
  - Research site021, Beijing, Beijing Municipality
  - Research site02, Beijing, Beijing Municipality
  - Research site01, Beijing, Beijing Municipality
  - Research site013, Beijing, Beijing Municipality
  - Research site010, Chongqing, Chongqing Municipality
  - Research site05, Xiamen, Fujian
  - Research site011, Shenzhen, Guangdong
  - Research site016, Nanning, Guangxi
  - Research site017, Shijiazhuang, Hebei
  - Research site018, Harbin, Heilongjiang
  - Research site04, Zhengzhou, Henan
  - Research site012, Changsha, Hunan
  - Research site015, Changchun, Jilin
  - Research site06, Shenyang, Liaoning
  - Research site07, Shenyang, Liaoning
  - Research site014, Hohhot, Neimenggu
  - Research site020, Xi’an, Shanxi
  - Research site03, Hubei, Wuhan
  - Research site019, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No